CLINICAL TRIAL: NCT01410058
Title: Effect of Moringa Oleifera (Moringa, Drumstick/Horseradish Tree) on The Pharmacokinetics of Efavirenz and Nevirapine In-vivo.
Brief Title: Moringa Oleifera- Antiretroviral Pharmacokinetic Drug Interaction
Status: Completed | Type: Observational
Sponsor: University of Zimbabwe (Other)
Collaborators: State University of New York at Buffalo (Other); Biomedical Research and Training Institute (Other)
Responsible Party: Principal Investigator, Tsitsi Grace Monera, Lecturer, University of Zimbabwe
Other Study IDs: MO 001
Record Dates: First submitted 2011-08-03; First posted 2011-08-04 (Estimated); Results first posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: HIV
Keywords: HIV; antiretroviral drug interaction; herbal medicine; pharmacokinetics; herbal pharmacology
MeSH Terms: interventions — flocculant protein MO 2.1, Moringa oleifera; efavirenz; Nevirapine; Tablets

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma, urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Nevirapine: HIV positive patients on nevirapine containing regimen, taking Moringa oleifera leaf powder
  Interventions: Dietary Supplement: Moringa oleifera; Drug: Nevirapine 200Mg Oral Tablet
- Efavirenz: HIV positive patients on efavirenz containing regimen, taking Moringa oleifera
  Interventions: Dietary Supplement: Moringa oleifera; Drug: Efavirenz 600mg

INTERVENTIONS:
Dietary Supplement: Moringa oleifera — leaf powder, 1.85g once daily, hard gelatin capsules
  Other Names: moringa; drumstick tree; horseradish tree
Drug: Efavirenz 600mg — Efavirenz 600mg based regimen
  Groups: Efavirenz
Drug: Nevirapine 200Mg Oral Tablet — Nevirapine 200mg based regimen
  Groups: Nevirapine

SUMMARY:
A study will be conducted by scientists from the University of Zimbabwe to determine if antiretroviral drugs are affected by taking herbs at the same time. This is important because herbal medicines may interact with modern medicine to increase or decrease the amount of medication in the body.

The drugs nevirapine and efavirenz will be studied. Both drugs are routinely used as part of combination therapy for treating HIV. In this study it will be determined whether the concentrations of the antiretroviral drugs nevirapine and efavirenz are low, high or are in the desired range when taken together with the herb moringa.

DETAILED DESCRIPTION:
The use of herbal supplements is widespread in Africa, particularly for the management of HIV and AIDS. In Zimbabwe, the prevalence of herbal medicine use in HIV-infected people is as high as 79% (Sebit et al., 2000). Several studies have shown that the herb Moringa oleifera is among the top 10 herbs most commonly used by HIV-positive people in Zimbabwe (Makomeya et al 2004, Monera et al 2008). Another review also cited Moringa as one of the 53 most important African medicinal plants presently traded (van den Bout-van den Beukel et al 2006). Others included Hypoxis hemerocallidea (African potato) and Sutherlandia frutescens-(Cancer bush). Moringa is rich in β-carotene, protein, vitamin C, calcium and potassium and act as a good source of natural antioxidants (Anwar et al.,2007).It is recommended by non-governmental organisations and some African governments as an immune booster and a nutritional supplement for people living with HIV and AIDS (Ncube, 2006). Most advocates and users believe that since the herb is natural, it is free from all side effects and interactions.

Concomitant use of herbs with conventional drugs may lead to herb-drug interactions in the same way that two or more co-administered drugs may interact. Herbal constituents that are substrates for the same enzymes or transporters of conventional drugs may induce or inhibit the enzymes and/or transporter activity. Pharmacokinetic endpoints such as area under the curve (AUC), time to maximum plasma concentration (tmax), peak plasma concentration (Cmax), trough concentration (Cmin), clearance (CL), volume of distribution (Vd/F) and half-life (T1/2) may be altered significantly resulting in toxicity, more severe adverse effects, sub-therapeutic drug concentrations, HIV resistance and treatment failure.The risk of interaction increases as the number of co-administered drugs increases (de Maat et al 2003). As a result, people taking herbal medicines while on antiretroviral therapy are at very high risk because of the multitude use of highly active antiretroviral drugs and treatment of opportunistic infections, and also because herbs contain a wide range of bioactive chemical constituents.

However, evidence based information of such effects is usually lacking and as such; health practitioners' ability to make relevant clinical decisions is limited. Results of a review of in vitro studies suggest a need for in vivo metabolic drug-drug interaction studies (van den Bout-van den Beukel et al 2006). Preliminary in vivo studies in animal models can serve as a basis for clinical trials, the results of which are considered the gold standard in this era of evidence-based medicine.

Primary objectives

1. To compare the steady-state pharmacokinetics of nevirapine and efavirenz in HIV-positive patients before and after supplementation with Moringa oleifera leaf powder
2. To compare the single dose pharmacokinetics of nevirapine and efavirenz in rat models before and after supplementation with Moringa oleifera leaf powder

   Secondary objectives
3. To determine the bioavailability of Moringa oleifera leaf powder in humans after oral dosing using beta carotene as a bio marker.
4. To compare urine chemistries and liver function tests in HIV patients before and after supplementation with Moringa oleifera leaf powder
5. To determine the presence of any genetic variation in the participants in the genes that code for CYP3A4 and CYP2B6

ELIGIBILITY:
Inclusion Criteria:

* HIV positive,
* ≥ 4 weeks on Nevirapine or , ≥ 2 weeks on Efavirenz containing regimen,
* Supplements HAART with Moringa oleifera.

Exclusion Criteria:

Known hepatic, intestinal or renal disease,smoking, chronic alcohol ingestion, poor venous access, chronic alcohol ingestion, pregnant, smoking, on rifampicin, ketoconazole, isoniazid, breastfeeding, anaemia,vomiting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV Opportunistic infections clinic
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2013-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tsitsi G Monera, BPharmHons, MPhil, MSc CT, Principal Investigator — University of Zimbabwe
Locations (1):
- Parirenyatwa Hospital OI Clinic, Harare, Zimbabwe

REFERENCES:
- [Background] Anwar F, Latif S, Ashraf M, Gilani AH. Moringa oleifera: a food plant with multiple medicinal uses. Phytother Res. 2007 Jan;21(1):17-25. doi: 10.1002/ptr.2023. PMID 17089328
- [Background] Sebit MB, Chandiwana SK, Latif AS, Gomo E, Acuda SW, Makoni F, Vushe J. Quality of life evaluation in patients with HIV-I infection: the impact of traditional medicine in Zimbabwe. Cent Afr J Med. 2000 Aug;46(8):208-13. PMID 11317592
- [Background] van den Bout-van den Beukel CJ, Koopmans PP, van der Ven AJ, De Smet PA, Burger DM. Possible drug-metabolism interactions of medicinal herbs with antiretroviral agents. Drug Metab Rev. 2006;38(3):477-514. doi: 10.1080/03602530600754065. PMID 16877262
- [Derived] Monera-Penduka TG, Maponga CC, Wolfe AR, Wiesner L, Morse GD, Nhachi CF. Effect of Moringa oleifera Lam. leaf powder on the pharmacokinetics of nevirapine in HIV-infected adults: a one sequence cross-over study. AIDS Res Ther. 2017 Mar 14;14:12. doi: 10.1186/s12981-017-0140-4. eCollection 2017. PMID 28293270
- [Derived] Monera-Penduka TG, Maponga CC, Morse GD, Nhachi CFB. Capacity for ethical and regulatory review of herbal trials in developing countries: a case study of Moringa oleifera research in HIV-infected patients. J Pharm Policy Pract. 2017 Feb 20;10:9. doi: 10.1186/s40545-017-0099-5. eCollection 2017. PMID 28250958

RESULTS

PARTICIPANT FLOW:
Recruitment Details: HIV-infected male and female adults reporting for routine HIV clinic visits at a referral hospital in Zimbabwe were identified through an interviewer-administered questionnaire.
Pre-assignment Details: The study had a minimum 3-week herbal medication wash out period prior to the first dosing to reduce the possibility of carryover from any type of previously used moringa or other herbal medication, so the participants would have the same baseline.
Groups:
- Efavirenz: HIV positive patients on efavirenz containing regimen, taking Moringa oleifera leaf powder
Period: Washout Day 0
Arm/Group | Nevirapine | Efavirenz
Started | 13 | 6
Completed | 13 | 6
Not Completed | 0 | 0
Period: Baseline Day 22
Arm/Group | Nevirapine | Efavirenz
Started | 13 | 6
Completed | 13 | 6
Not Completed | 0 | 0
Period: Day 35
Arm/Group | Nevirapine | Efavirenz
Started | 13 | 6
Completed | 13 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 11/13 were analysed in the nevirapine arm. 2 had missing data due to insufficient blood sample and were excluded from analysis.
  6/6 were analysed for efavirenz arm
Groups:
- Nevirapine: HIV positive patients on nevirapine containing regimen, taking Moringa oleifera leaf powder
  Moringa oleifera: leaf powder, 1.85g once daily as hard gelatin capsules
- Efavirenz: HIV positive patients on efavirenz containing regimen, taking Moringa oleifera
  Moringa oleifera: leaf powder, 1.85g once daily as hard gelatin capsules
- Total: Total of all reporting groups
Arm/Group | Nevirapine | Efavirenz | Total
Number analyzed (Participants) | 11 | 6 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (8) | 43 (8) | 44 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 3 | 2 | 5
Weight [Mean (Standard Deviation); unit: kg] | 63.5 (7.5) | 72.5 (17.0) | 65.9 (12.0)

OUTCOME MEASURES:

1. Primary Outcome: AUC
Description: Area under the plasma concentration time curve, determined using a non-compartmental approach by means of the Phoenix WinNonlin software application. Time points for sample collection were 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 h
Time Frame: Baseline (day 22), Post-moringa (day 35)
Population: Only participants with complete data were included
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*microgram/mL
Groups:
- Nevirapine: HIV positive patients on nevirapine containing regimen, taking Moringa oleifera leaf powder
  Moringa oleifera: leaf powder
- Efavirenz: HIV positive patients on efavirenz containing regimen, taking Moringa oleifera
  Moringa oleifera: leaf powder
Arm/Group | Nevirapine | Efavirenz
Number analyzed (Participants) | 11 | 6
h*microgram/mL
  Baseline (Day 22) | 94.17 (25.24) | 34.67 (24.85)
  Post-moringa (Day 35) | 100.44 (27.65) | 32.58 (38.75)

2. Secondary Outcome: C12h
Description: plasma concentration 12h post dose, determined using a non-compartmental approach by means of the Phoenix WinNonlin software application. Time points for sample collection were 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 h
Time Frame: Baseline (Day 22); Post-moringa (Day 35)
Population: Only patients with complete data were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/mL
Arm/Group | Nevirapine | Efavirenz
Number analyzed (Participants) | 11 | 6
microgram/mL
  Baseline (Day 22) | 7.30 (25.85) | 2.96 (18.75)
  Post-moringa (Day 35) | 7.55 (28.56) | 2.53 (21.35)

3. Other Pre Specified Outcome: Cmax
Description: Maximum plasma concentration post does, determined using a non-compartmental approach by means of the Phoenix WinNonlin software application. Time points for sample collection were 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 h
Time Frame: Baseline (day 22), Post-moringa (day 35)
Population: Only patients with complete data were included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/mL
Arm/Group | Nevirapine | Efavirenz
Number analyzed (Participants) | 11 | 6
microgram/mL
  Baseline (Day 22) | 9.92 (26.93) | 5.08 (22.95)
  Post-moringa (Day 35) | 10.57 (29.62) | 5.51 (38.28)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at baseline (day 22) and at final visit (day 35).
Description: All participants were monitored for adverse events throughout the study. The study medical officer documented any adverse events observed from clinical examinations or self-reported by the participants at each of the two visits. Urinalysis and Serum biochemistries were determined and graded based on CTCAE.
Arm/Group | Nevirapine | Efavirenz
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/6
Other Adverse Events (participants affected / at risk) | 4/13 | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nevirapine (N=13) | Efavirenz (N=6)
Altered creatinine clearance (Renal and urinary disorders) | 0 (0) | 2 (2) — Creatinine clearance outside range 88-137 mL/min
Elevated liver transaminase (Hepatobiliary disorders) | 4 (5) | 4 (4) — greater than upper limit of normal - 3 times upper limit of normal

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No